CLINICAL TRIAL: NCT01275170
Title: A Single-Dose Study to Investigate the Pharmacokinetics of MK-7655 in Subjects With Impaired Renal Function
Brief Title: A Single-Dose Study to Investigate the Pharmacokinetics of MK-7655 in Participants With Impaired Renal Function (MK-7655-005)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7655-005
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Infectious Disease
MeSH Terms: conditions — Communicable Diseases | interventions — relebactam; Cilastatin, Imipenem Drug Combination; Caffeine; Midazolam; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Panel A Mild Renal Impairment (Experimental): Participants with an eGFR of >50 to <80 mL/min/1.73 m^2 receive a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV in Part 1.
  Interventions: Drug: MK-7655; Drug: Imipenem + Cilastatin
- Panel B Healthy Participants (Experimental): A subset of healthy control participants were matched specifically to participants in Panel A and receive a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV in Part 1.
  Interventions: Drug: MK-7655; Drug: Imipenem + Cilastatin
- Panel C Moderate Renal Impairment (Experimental): Participants with an eGFR of 30 to 50 mL/min/1.73 m^2 receive a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV in Part 1.
  Interventions: Drug: MK-7655; Drug: Imipenem + Cilastatin
- Panel D Healthy Participants (Experimental): A subset of healthy control participants were matched specifically to participants in Panel C and receive a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV in Part 1.
  Interventions: Drug: MK-7655; Drug: Imipenem + Cilastatin
- Panel E Severe Renal Impairment (Experimental): Participants with an eGFR <30 mL/min/1.73 m^2 receive a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV in Part 1. In Part 2, participants receive an oral cocktail containing caffeine 200 mg, midazolam 2 mg, and omeprazole 40 mg.
  Interventions: Drug: MK-7655; Drug: Imipenem + Cilastatin; Drug: Caffeine; Drug: Midazolam; Drug: Omeprazole
- Panel F Healthy Participants (Experimental): A subset of healthy control participants were matched specifically to participants in Panel E and receive a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV in Part 1. In Part 2, participants receive an oral cocktail containing caffeine 200 mg, midazolam 2 mg, and omeprazole 40 mg.
  Interventions: Drug: MK-7655; Drug: Imipenem + Cilastatin; Drug: Caffeine; Drug: Midazolam; Drug: Omeprazole
- Panel G End Stage Renal Disease with Hemodialysis (ESRD/HD) (Experimental): Participants with ESRD/HD receive a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV postdialysis (Part 1, Period 1) and predialysis (Part 1, Period 2). In Part 2, participants receive an oral cocktail containing caffeine 200 mg, midazolam 2 mg, and omeprazole 40 mg predialysis (Part 2, Period 1) and postdialysis (Part 2, Period 2).
  Interventions: Drug: MK-7655; Drug: Imipenem + Cilastatin; Drug: Caffeine; Drug: Midazolam; Drug: Omeprazole
- Panel H Healthy Volunteers (Experimental): A subset of healthy control participants were matched specifically to participants in Panel G and receive a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV in Part 1. In Part 2, participants receive an oral cocktail containing caffeine 200 mg, midazolam 2 mg, and omeprazole 40 mg.
  Interventions: Drug: MK-7655; Drug: Imipenem + Cilastatin; Drug: Caffeine; Drug: Midazolam; Drug: Omeprazole

INTERVENTIONS:
Drug: MK-7655 — 125 mg intravenous (IV) over 30 minutes as a single dose
  Other Names: RELEBACTAM®
Drug: Imipenem + Cilastatin — 250 mg IV over 30 minutes as a single dose
  Other Names: PRIMAXIN®
Drug: Caffeine — Caffeine caplet, single 200 mg dose, orally
  Other Names: No Doz®
  Arms: Panel E Severe Renal Impairment; Panel F Healthy Participants; Panel G End Stage Renal Disease with Hemodialysis (ESRD/HD); Panel H Healthy Volunteers
Drug: Midazolam — Midazolam hcl syrup single 2.0 mg dose by mouth.
  Other Names: VERSED®
  Arms: Panel E Severe Renal Impairment; Panel F Healthy Participants; Panel G End Stage Renal Disease with Hemodialysis (ESRD/HD); Panel H Healthy Volunteers
Drug: Omeprazole — Omeprazole tablets, single 40 mg dose (as two 20 mg tablets), orally
  Other Names: PRILOSEC®
  Arms: Panel E Severe Renal Impairment; Panel F Healthy Participants; Panel G End Stage Renal Disease with Hemodialysis (ESRD/HD); Panel H Healthy Volunteers

SUMMARY:
This is a 2-part study of the pharmacokinetics (PK) of MK-7655. In Part I, the PK of a single 125 mg dose of MK-7655 given in combination with 250 mg of PRIMAXIN® (imipenem + cilastatin) will be determined in participants with impaired renal function and matched control participants. In Part II, the potential for renal insufficiency to affect non-renal clearance mechanisms will be investigated.

ELIGIBILITY:
Inclusion criteria

* Participants of reproductive potential (male or female) must be willing to use contraception.
* Body Mass Index (BMI) ≤40 kg/m^2
* Weight >60 kg at screening visit
* No clinically significant abnormality on electrocardiogram (ECG) at screening visit and/or prior to administration of the initial dose of study drug
* Panels A-D: smokers will be limited to no more that 10 cigarettes per day.
* Panels E-H: nonsmoker or has not used nicotine for at least 6 months
* In good health (stable health for participants with renal impairment)

Exclusion criteria

* Pregnant or breastfeeding.
* History of recent stroke, chronic seizures, or major neurological disorder
* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, immunological, respiratory, or genitourinary abnormalities or diseases
* History of malignant neoplastic disease. Exceptions: (1) adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix; (2) other malignancies that have been successfully treated ≥10 years prior to the screening visit
* Panels A-D: Use of any medication (prescription or non-prescription) or herbal remedies (such as St. John's Wort [Hypericum perforatum]) beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of study drug to the post study visit
* Panels E-H: Use of any medication (prescription or non-prescription) or herbal remedies (such as St. John's Wort [Hypericum perforatum]) that are inhibitors or inducers of CYP1A2, CYP2C19, CYP34A, or substrates of CYP2C19, beginning approximately 2 weeks (or 5 half-lives) prior to administration of the probe cocktail, until the post-study visit
* Consumption of greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL/10 ounces], wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]) per day
* Consumption of greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, or other caffeinated beverages per day
* Major surgery, donation or loss of 1 unit of blood (approximately 500 mL), or participation in another investigational study within 4 weeks prior to the screening visit
* History of multiple and/or severe allergies (including latex allergy), or prior anaphylactic reaction or intolerability to prescription or non-prescription drugs or food
* History of hypersensitivity to PRIMAXIN® IV or other beta lactam antibiotic (including but not limited to penicillins, cephalosporins, monobactams and carbapenems)
* Regular user (including recreational use of drugs [including alcohol]) within approximately 12 months of screening visit
* History of kidney removal and/or renal transplant
* History of Clostridium difficile colitis or known C. difficile colonization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-01-28 (Actual); Primary Completion 2012-03-05 (Actual); Study Completion 2012-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Bhagunde P, Colon-Gonzalez F, Liu Y, Wu J, Xu SS, Garrett G, Jumes P, Lasseter K, Marbury T, Rizk ML, Lala M, Rhee EG, Butterton JR, Boundy K. Impact of renal impairment and human organic anion transporter inhibition on pharmacokinetics, safety and tolerability of relebactam combined with imipenem and cilastatin. Br J Clin Pharmacol. 2020 May;86(5):944-957. doi: 10.1111/bcp.14204. Epub 2020 Jan 23. PMID 31856304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with varying degrees of renal impairment, or with end-stage renal disease (ESRD) requiring hemodialysis (HD) [based on estimated glomerular filtration rate (eGFR)], or healthy matched controls were enrolled at 2 study sites in the United States.
Pre-assignment Details: All panels participated in Part 1 of the study. Panels E to H also participated in Part 2 of the study.
Groups:
- Panel A: Mild Renal Impairment: Participants with an eGFR of >50 to <80 mL/min/1.73m² receive a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV in Part 1.
- Panel B: Healthy Controls to Panel A: Healthy control participants were matched specifically to participants in Panel A and received a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV in Part 1.
- Panel C: Moderate Renal Impairment: Participants with an eGFR of 30 to 50 mL/min/1.73m² receive a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV in Part 1.
- Panel D: Healthy Controls to Panel C: Healthy control participants were matched specifically to participants in Panel C and received a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV in Part 1.
- Panel E: Severe Renal Impairment: Participants with an eGFR <30 mL/min/1.73m² receive a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV in Part 1. In Part 2, participants receive an oral cocktail containing caffeine 200 mg, midazolam 2 mg, and omeprazole 40 mg.
- Panel F: Healthy Controls to Panel E: A subset of healthy control participants was matched specifically to participants in Panel E and received a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV in Part 1.
- Panel G: ESRD/HD Participants: Participants with ESRD/HD receive a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV postdialysis (Part 1, Period 1) and predialysis (Part 1, Period 2). In Part 2, participants receive an oral cocktail containing caffeine 200 mg, midazolam 2 mg, and omeprazole 40 mg predialysis (Part 2, Period 1) and postdialysis (Part 2, Period 2).
- Panel H: Healthy Controls to Panel G: Healthy control participants were matched specifically to participants in Panel G and received a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV in Part 1.
Period: Part 1: Period 1
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Participants | Panel H: Healthy Controls to Panel G
Started (Randomized) | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Treated | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Equipment malfunction before study drug | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Period 2
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Participants | Panel H: Healthy Controls to Panel G
Started | 0 (Panel A participated in Part 1, Period 1 only.) | 0 (Panel B participated in Part 1, Period 1 only.) | 0 (Panel C participated in Part 1, Period 1 only.) | 0 (Panel D participated in Part 1, Period 1 only.) | 0 (Panel E participated in Part 1, Period 1 and Part 2, Period 1.) | 0 (Panel E participated in Part 1, Period 1 and Part 2, Period 1.) | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Period 1
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Participants | Panel H: Healthy Controls to Panel G
Started | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Period 2
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Participants | Panel H: Healthy Controls to Panel G
Started | 0 | 0 | 0 | 0 | 0 (Panel E participated in Part 1, Period 1 and Part 2, Period 1.) | 0 (Panel F participated in Part 1, Period 1 and Part 2, Period 1.) | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Base Population consists of 49 randomized participants, including n=1 participant in Panel A who was discontinued prior to receiving study drug due to an equipment malfunction.
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Participants | Panel H: Healthy Controls to Panel G | Total
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.1 (3.4) | 64.5 (3.9) | 68.3 (5.0) | 64.2 (5.7) | 62.8 (7.5) | 60.5 (6.4) | 44.5 (7.9) | 41.5 (11.5) | 59.9 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 3 | 3 | 3 | 2 | 2 | 21
  Male | 4 | 4 | 3 | 3 | 3 | 3 | 4 | 4 | 28

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Area Under the Plasma Concentration-time Curve From Dosing to Infinity (AUC0-inf) of MK-7655 in Combination With PRIMAXIN®
Description: AUC0-∞ is a measure of the mean (extrapolated) plasma drug concentration after dosing to infinity.
Time Frame: Predose and 0.08, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, and 14 hours postdose
Population: Treated participants who complied with the protocol sufficiently to ensure that generated data were likely to exhibit the effects of treatment, according to the underlying scientific model, are included. Per protocol, data for Panel G were reported separately for post-dialysis and pre-dialysis.
Measure: Geometric Mean (95% Confidence Interval); unit: µM*hr
Groups:
- Panel E: Severe Renal Impairment: Participants with an eGFR <30 mL/min/1.73m² receive a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV in Part 1.
- Panel G: ESRD/HD Period 1 Postdialysis; Panel G: ESRD/HD Period 2 Predialysis: Participants with ESRD/HD receive a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV postdialysis (Part 1, Period 1) and predialysis (Part 1, Period 2).
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel H: Healthy Controls to Panel G | Panel G: ESRD/HD Period 2 Predialysis
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
µM*hr | 73.5 [50.0 to 108] | 45.0 [32.4 to 62.6] | 115 [79.8 to 165] | 52.3 [37.7 to 72.7] | 236 [171 to 325] | 48.5 [35.3 to 66.4] | 414 [280 to 612] | 44.5 [29.1 to 67.9] | 78.0 [50.3 to 121]
Statistical Analysis 1: Comparison: Panel A: Mild Renal Impairment vs Panel B: Healthy Controls to Panel A; Test type: Other — Geometric mean ratio (GMR) [Renal Impairment/Healthy Control]; GMR = 1.63, 90% CI 2-sided [1.12 to 2.39]
Statistical Analysis 2: Comparison: Panel C: Moderate Renal Impairment vs Panel D: Healthy Controls to Panel C; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 2.19, 90% CI 2-sided [1.51 to 3.18]
Statistical Analysis 3: Comparison: Panel E: Severe Renal Impairment vs Panel F: Healthy Controls to Panel E; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 4.87, 90% CI 2-sided [3.37 to 7.04]
Statistical Analysis 4: Comparison: Panel G: ESRD/HD Period 1 Postdialysis vs Panel H: Healthy Controls to Panel G; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 9.32, 90% CI 2-sided [6.45 to 13.46]
Statistical Analysis 5: Comparison: Panel H: Healthy Controls to Panel G vs Panel G: ESRD/HD Period 2 Predialysis; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 1.76, 90% CI 2-sided [1.20 to 2.58]

2. Secondary Outcome: Part 1: Concentration at End of Infusion (Ceoi) of MK-7655 in Combination With PRIMAXIN®
Description: Ceoi is the observed plasma drug concentration at the end of IV infusion.
Time Frame: At 0.5 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µM
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel H: Healthy Controls to Panel G | Panel G: ESRD/HD Period 2 Predialysis
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
µM | 22.4 [13.0 to 38.7] | 20.4 [12.8 to 32.7] | 23.5 [14.0 to 39.4] | 22.5 [14.1 to 35.9] | 23.6 [15.0 to 37.2] | 18.1 [11.6 to 28.4] | 53.1 [30.7 to 91.9] | 22.7 [12.5 to 41.0] | 19.3 [11.2 to 33.4]
Statistical Analysis 1: Comparison: Panel A: Mild Renal Impairment vs Panel B: Healthy Controls to Panel A; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 1.10, 90% CI 2-sided [0.64 to 1.88]
Statistical Analysis 2: Comparison: Panel C: Moderate Renal Impairment vs Panel D: Healthy Controls to Panel C; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 1.04, 90% CI 2-sided [0.62 to 1.77]
Statistical Analysis 3: Comparison: Panel E: Severe Renal Impairment vs Panel F: Healthy Controls to Panel E; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 1.30, 90% CI 2-sided [0.77 to 2.20]
Statistical Analysis 4: Comparison: Panel G: ESRD/HD Period 1 Postdialysis vs Panel H: Healthy Controls to Panel G; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 2.34, 90% CI 2-sided [1.39 to 3.96]
Statistical Analysis 5: Comparison: Panel H: Healthy Controls to Panel G vs Panel G: ESRD/HD Period 2 Predialysis; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.85, 90% CI 2-sided [0.50 to 1.44]

3. Secondary Outcome: Part 1: Predicted Clearance (CLpred) of MK-7655 in Combination With PRIMAXIN®
Description: CLpred is the predicted apparent total body clearance of drug.
Time Frame: Predose and 0.08, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, and 14 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mL/min
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel H: Healthy Controls to Panel G | Panel G: ESRD/HD Period 2 Predialysis
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
mL/min | 81.3 [55.3 to 119] | 133 [95.5 to 185] | 52.1 [36.2 to 74.9] | 114 [82.3 to 159] | 25.3 [18.4 to 34.9] | 123 [90.0 to 169] | 14.4 [9.77 to 21.3] | 135 [88.1 to 206] | 76.6 [49.4 to 119]
Statistical Analysis 1: Comparison: Panel A: Mild Renal Impairment vs Panel B: Healthy Controls to Panel A; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.61, 90% CI 2-sided [0.42 to 0.90]
Statistical Analysis 2: Comparison: Panel C: Moderate Renal Impairment vs Panel D: Healthy Controls to Panel C; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.46, 90% CI 2-sided [0.31 to 0.66]
Statistical Analysis 3: Comparison: Panel E: Severe Renal Impairment vs Panel F: Healthy Controls to Panel E; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.21, 90% CI 2-sided [0.14 to 0.30]
Statistical Analysis 4: Comparison: Panel G: ESRD/HD Period 1 Postdialysis vs Panel H: Healthy Controls to Panel G; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.11, 90% CI 2-sided [0.07 to 0.16]
Statistical Analysis 5: Comparison: Panel H: Healthy Controls to Panel G vs Panel G: ESRD/HD Period 2 Predialysis; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.57, 90% CI 2-sided [0.39 to 0.84]

4. Secondary Outcome: Part 1: Predicted Volume of Distribution During the Terminal Phase (VZpred) of MK-7655 in Combination With PRIMAXIN®
Description: VZpred is the predicted volume of distribution during the terminal phase.
Time Frame: Predose and 0.08, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, and 14 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: liters (L)
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel H: Healthy Controls to Panel G | Panel G: ESRD/HD Period 2 Predialysis
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
liters (L) | 21.4 [17.6 to 26.1] | 21.6 [18.2 to 25.5] | 22.2 [18.4 to 26.7] | 21.9 [18.5 to 25.9] | 20.1 [17.1 to 23.7] | 22.4 [19.0 to 26.3] | 16.2 [13.3 to 19.8] | 17.0 [13.6 to 21.1] | 55.7 [44.5 to 69.7]
Statistical Analysis 1: Comparison: Panel A: Mild Renal Impairment vs Panel B: Healthy Controls to Panel A; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.99, 90% CI 2-sided [0.82 to 1.21]
Statistical Analysis 2: Comparison: Panel C: Moderate Renal Impairment vs Panel D: Healthy Controls to Panel C; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 1.01, 90% CI 2-sided [0.84 to 1.22]
Statistical Analysis 3: Comparison: Panel E: Severe Renal Impairment vs Panel F: Healthy Controls to Panel E; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.90, 90% CI 2-sided [0.74 to 1.08]
Statistical Analysis 4: Comparison: Panel G: ESRD/HD Period 1 Postdialysis vs Panel H: Healthy Controls to Panel G; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.96, 90% CI 2-sided [0.79 to 1.16]
Statistical Analysis 5: Comparison: Panel H: Healthy Controls to Panel G vs Panel G: ESRD/HD Period 2 Predialysis; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 3.28, 90% CI 2-sided [2.70 to 4.00]

5. Secondary Outcome: Part 1: Time of Maximum Plasma Concentration (Tmax) of MK-7655 in Combination With PRIMAXIN®
Description: Tmax is the time at which the highest plasma drug concentration was observed.
Time Frame: Predose and 0.08, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, and 14 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel H: Healthy Controls to Panel G | Panel G: ESRD/HD Period 2 Predialysis
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 0.50 [0.48 to 1.27] | 0.50 [0.48 to 0.52] | 0.50 [0.48 to 0.75] | 0.49 [0.48 to 0.75] | 0.48 [0.48 to 1.00] | 0.48 [0.48 to 0.75] | 0.48 [0.08 to 1.00] | 0.48 [0.48 to 0.48] | 0.48 [0.48 to 0.55]

6. Secondary Outcome: Part 1: Apparent Plasma Half-life (t½) of MK-7655 in Combination With PRIMAXIN®
Description: Apparent t½ is the amount of time for the maximum drug concentration to decrease by 50%.
Time Frame: Predose and 0.08, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, and 14 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel H: Healthy Controls to Panel G | Panel G: ESRD/HD Period 2 Predialysis
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 2.63 (26.4) | 1.75 (16.6) | 4.51 (25.7) | 2.10 (31.0) | 8.65 (31.0) | 2.00 (10.4) | 15.6 (103.1) | 1.79 (13.9) | 10.5 (100.6)

7. Secondary Outcome: Part 1: AUC0-inf of Imipenem in Combination With MK-7655
Description: Imipenem is 1 of the 2 constituents of PRIMAXIN®. AUC0-∞ is a measure of the mean (extrapolated) plasma drug concentration after dosing to infinity.
Time Frame: Predose and 0.08, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, and 14 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel H: Healthy Controls to Panel G | Panel G: ESRD/HD Period 2 Predialysis
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
µM*hr | 77.3 [58.9 to 101] | 55.0 [43.5 to 69.5] | 101 [77.9 to 130] | 66.0 [52.2 to 83.3] | 160 [127 to 201] | 63.8 [51.0 to 79.9] | 223 [169 to 293] | 71.8 [53.4 to 96.5] | 71.2 [54.2 to 93.6]
Statistical Analysis 1: Comparison: Panel A: Mild Renal Impairment vs Panel B: Healthy Controls to Panel A; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 1.41, 90% CI 2-sided [1.07 to 1.84]
Statistical Analysis 2: Comparison: Panel C: Moderate Renal Impairment vs Panel D: Healthy Controls to Panel C; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 1.53, 90% CI 2-sided [1.17 to 1.99]
Statistical Analysis 3: Comparison: Panel E: Severe Renal Impairment vs Panel F: Healthy Controls to Panel E; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 2.51, 90% CI 2-sided [1.93 to 3.26]
Statistical Analysis 4: Comparison: Panel G: ESRD/HD Period 1 Postdialysis vs Panel H: Healthy Controls to Panel G; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 3.10, 90% CI 2-sided [2.39 to 4.03]
Statistical Analysis 5: Comparison: Panel H: Healthy Controls to Panel G vs Panel G: ESRD/HD Period 2 Predialysis; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.99, 90% CI 2-sided [0.76 to 1.29]

8. Secondary Outcome: Part 1: Ceoi of Imipenem in Combination With MK-7655
Description: Imipenem is 1 of the 2 constituents of PRIMAXIN®. Ceoi is the observed plasma drug concentration at the end of IV infusion.
Time Frame: At 0.5 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µM
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel H: Healthy Controls to Panel G | Panel G: ESRD/HD Period 2 Predialysis
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6
µM | 40.7 [22.7 to 73.2] | 35.3 [21.3 to 58.5] | 45.6 [26.2 to 79.5] | 42.6 [25.8 to 70.4] | 46.9 [28.7 to 76.5] | 35.5 [21.9 to 57.6] | 103 [57.1 to 186] | 41.8 [22.1 to 79.1] | 35.9 [19.9 to 64.7]
Statistical Analysis 1: Comparison: Panel A: Mild Renal Impairment vs Panel B: Healthy Controls to Panel A; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 1.15, 90% CI 2-sided [0.65 to 2.06]
Statistical Analysis 2: Comparison: Panel C: Moderate Renal Impairment vs Panel D: Healthy Controls to Panel C; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 1.07, 90% CI 2-sided [0.61 to 1.89]
Statistical Analysis 3: Comparison: Panel E: Severe Renal Impairment vs Panel F: Healthy Controls to Panel E; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 1.32, 90% CI 2-sided [0.75 to 2.32]
Statistical Analysis 4: Comparison: Panel G: ESRD/HD Period 1 Postdialysis vs Panel H: Healthy Controls to Panel G; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 2.46, 90% CI 2-sided [1.40 to 4.33]
Statistical Analysis 5: Comparison: Panel H: Healthy Controls to Panel G vs Panel G: ESRD/HD Period 2 Predialysis; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.86, 90% CI 2-sided [0.49 to 1.51]

9. Secondary Outcome: Part 1: CLpred of Imipenem in Combination With MK-7655
Description: Imipenem is 1 of the 2 constituents of PRIMAXIN®. CLpred is the predicted apparent total body clearance of drug.
Time Frame: Predose and 0.08, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, and 14 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mL/min
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel H: Healthy Controls to Panel G | Panel G: ESRD/HD Period 2 Predialysis
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
mL/min | 180 [137 to 236] | 253 [200 to 320] | 138 [107 to 179] | 211 [167 to 266] | 87.0 [69.4 to 109] | 218 [174 to 273] | 62.5 [47.5 to 82.1] | 194 [144 to 261] | 195 [149 to 257]
Statistical Analysis 1: Comparison: Panel A: Mild Renal Impairment vs Panel B: Healthy Controls to Panel A; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.71, 90% CI 2-sided [0.54 to 0.93]
Statistical Analysis 2: Comparison: Panel C: Moderate Renal Impairment vs Panel D: Healthy Controls to Panel C; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.65, 90% CI 2-sided [0.50 to 0.85]
Statistical Analysis 3: Comparison: Panel E: Severe Renal Impairment vs Panel F: Healthy Controls to Panel E; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.40, 90% CI 2-sided [0.31 to 0.52]
Statistical Analysis 4: Comparison: Panel G: ESRD/HD Period 1 Postdialysis vs Panel H: Healthy Controls to Panel G; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.32, 90% CI 2-sided [0.25 to 0.42]
Statistical Analysis 5: Comparison: Panel H: Healthy Controls to Panel G vs Panel G: ESRD/HD Period 2 Predialysis; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 1.01, 90% CI 2-sided [0.78 to 1.31]

10. Secondary Outcome: Part 1: VZpred of Imipenem in Combination With MK-7655
Description: Imipenem is 1 of the 2 constituents of PRIMAXIN®. VZpred is the predicted volume of distribution during the terminal phase.
Time Frame: Predose and 0.08, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, and 14 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: liters (L)
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel H: Healthy Controls to Panel G | Panel G: ESRD/HD Period 2 Predialysis
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
liters (L) | 21.1 [15.8 to 28.2] | 26.1 [20.4 to 33.5] | 22.3 [17.0 to 29.3] | 23.4 [18.3 to 30.0] | 20.0 [15.7 to 25.4] | 24.8 [19.6 to 31.5] | 20.5 [15.4 to 27.4] | 24.9 [18.2 to 34.1] | 63.3 [47.3 to 84.6]
Statistical Analysis 1: Comparison: Panel A: Mild Renal Impairment vs Panel B: Healthy Controls to Panel A; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.81, 90% CI 2-sided [0.61 to 1.08]
Statistical Analysis 2: Comparison: Panel C: Moderate Renal Impairment vs Panel D: Healthy Controls to Panel C; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.95, 90% CI 2-sided [0.72 to 1.26]
Statistical Analysis 3: Comparison: Panel E: Severe Renal Impairment vs Panel F: Healthy Controls to Panel E; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.80, 90% CI 2-sided [0.61 to 1.06]
Statistical Analysis 4: Comparison: Panel G: ESRD/HD Period 1 Postdialysis vs Panel H: Healthy Controls to Panel G; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.83, 90% CI 2-sided [0.63 to 1.09]
Statistical Analysis 5: Comparison: Panel H: Healthy Controls to Panel G vs Panel G: ESRD/HD Period 2 Predialysis; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 2.54, 90% CI 2-sided [1.93 to 3.36]

11. Secondary Outcome: Part 1: Tmax of Imipenem in Combination With MK-7655
Description: Tmax is the time at which the highest plasma drug concentration was observed.
Time Frame: Predose and 0.08, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, and 14 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel H: Healthy Controls to Panel G | Panel G: ESRD/HD Period 2 Predialysis
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 0.50 [0.48 to 0.82] | 0.50 [0.48 to 0.52] | 0.49 [0.48 to 0.50] | 0.48 [0.48 to 0.52] | 0.48 [0.48 to 1.00] | 0.48 [0.48 to 0.75] | 0.48 [0.08 to 0.48] | 0.48 [0.48 to 0.48] | 0.48 [0.48 to 0.55]

12. Secondary Outcome: Part 1: Apparent t½ of Imipenem in Combination With MK-7655
Description: Imipenem is 1 of the 2 constituents of PRIMAXIN®. Apparent t½ is the amount of time for the maximum drug concentration to decrease by 50%.
Time Frame: Predose and 0.08, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, and 14 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel H: Healthy Controls to Panel G | Panel G: ESRD/HD Period 2 Predialysis
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 1.54 (15.2) | 1.24 (10.8) | 2.18 (12.8) | 1.40 (21.1) | 2.78 (11.9) | 1.32 (5.8) | 3.24 (18.7) | 1.21 (13.7) | 3.20 (47.8)

13. Secondary Outcome: Part 1: AUC0-inf of Cilastin in Combination With MK-7655
Description: Cilastin is 1 of the 2 constituents of PRIMAXIN®. AUC0-∞ is a measure of the mean (extrapolated) plasma drug concentration after dosing to infinity.
Time Frame: Predose and 0.08, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, and 14 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel H: Healthy Controls to Panel G | Panel G: ESRD/HD Period 2 Predialysis
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
µM*hr | 71.7 [45.8 to 112] | 44.8 [30.5 to 65.9] | 100.0 [65.4 to 153] | 53.6 [36.6 to 78.6] | 300 [207 to 436] | 53.7 [37.2 to 77.6] | 777 [493 to 1220] | 56.5 [34.5 to 92.6] | 205 [123 to 343]
Statistical Analysis 1: Comparison: Panel A: Mild Renal Impairment vs Panel B: Healthy Controls to Panel A; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 1.60, 90% CI 2-sided [1.03 to 2.49]
Statistical Analysis 2: Comparison: Panel C: Moderate Renal Impairment vs Panel D: Healthy Controls to Panel C; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 1.86, 90% CI 2-sided [1.21 to 2.87]
Statistical Analysis 3: Comparison: Panel E: Severe Renal Impairment vs Panel F: Healthy Controls to Panel E; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 5.60, 90% CI 2-sided [3.64 to 8.59]
Statistical Analysis 4: Comparison: Panel G: ESRD/HD Period 1 Postdialysis vs Panel H: Healthy Controls to Panel G; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 13.75, 90% CI 2-sided [8.96 to 21.12]
Statistical Analysis 5: Comparison: Panel H: Healthy Controls to Panel G vs Panel G: ESRD/HD Period 2 Predialysis; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 3.64, 90% CI 2-sided [2.32 to 5.69]

14. Secondary Outcome: Part 1: Ceoi of Cilastin in Combination With MK-7655
Description: Cilastin is 1 of the 2 constituents of PRIMAXIN®. Ceoi is the observed plasma drug concentration at the end of IV infusion.
Time Frame: At 0.5 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µM
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel H: Healthy Controls to Panel G | Panel G: ESRD/HD Period 2 Predialysis
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6
µM | 43.4 [25.9 to 72.7] | 34.8 [22.3 to 54.4] | 48.7 [29.8 to 79.4] | 42.9 [27.5 to 66.8] | 53.3 [34.6 to 82.0] | 35.8 [23.4 to 54.8] | 111 [65.9 to 186] | 44.5 [25.4 to 78.0] | 41.7 [24.8 to 70.0]
Statistical Analysis 1: Comparison: Panel A: Mild Renal Impairment vs Panel B: Healthy Controls to Panel A; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 1.25, 90% CI 2-sided [0.75 to 2.08]
Statistical Analysis 2: Comparison: Panel C: Moderate Renal Impairment vs Panel D: Healthy Controls to Panel C; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 1.13, 90% CI 2-sided [0.69 to 1.87]
Statistical Analysis 3: Comparison: Panel E: Severe Renal Impairment vs Panel F: Healthy Controls to Panel E; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 1.49, 90% CI 2-sided [0.90 to 2.44]
Statistical Analysis 4: Comparison: Panel G: ESRD/HD Period 1 Postdialysis vs Panel H: Healthy Controls to Panel G; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 2.49, 90% CI 2-sided [1.51 to 4.09]
Statistical Analysis 5: Comparison: Panel H: Healthy Controls to Panel G vs Panel G: ESRD/HD Period 2 Predialysis; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.94, 90% CI 2-sided [0.57 to 1.54]

15. Secondary Outcome: Part 1: CLpred of Cilastin in Combination With MK-7655
Description: Cilastin is 1 of the 2 constituents of PRIMAXIN®. CLpred is the predicted apparent total body clearance of drug.
Time Frame: Predose and 0.08, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, and 14 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mL/min
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel H: Healthy Controls to Panel G | Panel G: ESRD/HD Period 2 Predialysis
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
mL/min | 162 [104 to 254] | 259 [176 to 381] | 116 [76.1 to 178] | 217 [148 to 318] | 38.7 [26.7 to 56.2] | 217 [150 to 313] | 15.0 [9.50 to 23.6] | 206 [126 to 337] | 56.6 [33.9 to 94.4]
Statistical Analysis 1: Comparison: Panel A: Mild Renal Impairment vs Panel B: Healthy Controls to Panel A; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.63, 90% CI 2-sided [0.40 to 0.97]
Statistical Analysis 2: Comparison: Panel C: Moderate Renal Impairment vs Panel D: Healthy Controls to Panel C; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.54, 90% CI 2-sided [0.35 to 0.83]
Statistical Analysis 3: Comparison: Panel E: Severe Renal Impairment vs Panel F: Healthy Controls to Panel E; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.18, 90% CI 2-sided [0.12 to 0.27]
Statistical Analysis 4: Comparison: Panel G: ESRD/HD Period 1 Postdialysis vs Panel H: Healthy Controls to Panel G; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.07, 90% CI 2-sided [0.05 to 0.11]
Statistical Analysis 5: Comparison: Panel H: Healthy Controls to Panel G vs Panel G: ESRD/HD Period 2 Predialysis; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.27, 90% CI 2-sided [0.18 to 0.43]

16. Secondary Outcome: Part 1: VZpred of Cilastin in Combination With MK-7655
Description: Cilastin is 1 of the 2 constituents of PRIMAXIN®. VZpred is the predicted volume of distribution during the terminal phase.
Time Frame: Predose and 0.08, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, and 14 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: liters (L)
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel H: Healthy Controls to Panel G | Panel G: ESRD/HD Period 2 Predialysis
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
liters (L) | 19.2 [14.8 to 24.9] | 23.9 [19.1 to 30.0] | 19.4 [15.2 to 24.9] | 21.4 [17.1 to 26.7] | 16.9 [13.6 to 21.0] | 21.2 [17.1 to 26.2] | 15.9 [12.2 to 20.7] | 21.0 [15.8 to 28.0] | 59.1 [43.9 to 79.6]
Statistical Analysis 1: Comparison: Panel A: Mild Renal Impairment vs Panel B: Healthy Controls to Panel A; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.80, 90% CI 2-sided [0.62 to 1.04]
Statistical Analysis 2: Comparison: Panel C: Moderate Renal Impairment vs Panel D: Healthy Controls to Panel C; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.91, 90% CI 2-sided [0.71 to 1.17]
Statistical Analysis 3: Comparison: Panel E: Severe Renal Impairment vs Panel F: Healthy Controls to Panel E; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.80, 90% CI 2-sided [0.62 to 1.03]
Statistical Analysis 4: Comparison: Panel G: ESRD/HD Period 1 Postdialysis vs Panel H: Healthy Controls to Panel G; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.76, 90% CI 2-sided [0.59 to 0.97]
Statistical Analysis 5: Comparison: Panel H: Healthy Controls to Panel G vs Panel G: ESRD/HD Period 2 Predialysis; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 2.81, 90% CI 2-sided [2.16 to 3.65]

17. Secondary Outcome: Part 1: Tmax of Cilastin in Combination With MK-7655
Description: Tmax is the time at which the highest plasma drug concentration was observed.
Time Frame: Predose and 0.08, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, and 14 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel H: Healthy Controls to Panel G | Panel G: ESRD/HD Period 2 Predialysis
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 0.50 [0.50 to 0.82] | 0.50 [0.48 to 0.52] | 0.49 [0.48 to 0.50] | 0.48 [0.48 to 0.52] | 0.48 [0.48 to 1.00] | 0.48 [0.48 to 0.48] | 0.48 [0.08 to 0.48] | 0.48 [0.48 to 0.48] | 0.48 [0.48 to 0.55]

18. Secondary Outcome: Part 1: Apparent t½ of Cilastin in Combination With MK-7655
Description: Cilastin is 1 of the 2 constituents of PRIMAXIN®. Apparent t½ is the amount of time for the maximum drug concentration to decrease by 50%.
Time Frame: Predose and 0.08, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, and 14 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel H: Healthy Controls to Panel G | Panel G: ESRD/HD Period 2 Predialysis
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 1.43 (31.9) | 1.08 (27.8) | 2.11 (20.5) | 1.19 (28.5) | 5.08 (59.2) | 1.09 (10.7) | 12.2 (118.5) | 1.14 (26.1) | 12.2 (131.5)

19. Secondary Outcome: Part 1: Renal Clearance (CLR) of MK-7655 in Urine
Description: CLR represents renal clearance in urine. Urine was collected for 24 hours postdose.
Time Frame: Predose to 24 hours postdose
Population: Treated participants with urine samples who complied with the protocol sufficiently to ensure that generated data were likely to exhibit the effects of treatment, according to the underlying scientific model, are included. Per protocol, Panel G was not sampled due to limitations in producing urine and was thus not included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel H: Healthy Controls to Panel G
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
mL/min | 69.8 (16.5) | 118 (19.8) | 38.4 (28.8) | 110 (36) | 22.3 (47.2) | 107 (20.9) | 110 (20)

20. Secondary Outcome: Part 1: CLR of Imipenem in Urine
Description: CLR represents renal clearance in urine. Urine was collected for 24 hours postdose.
Time Frame: Predose to 24 hours postdose
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel H: Healthy Controls to Panel G
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
mL/min | 75.0 (14.6) | 115 (18.4) | 41.1 (23.8) | 109 (29.2) | 17.4 (44.7) | 104 (10.5) | 99.1 (22.3)

21. Secondary Outcome: Part 1: CLR of Cilastin in Urine
Description: CLR represents renal clearance in urine. Urine was collected for 24 hours postdose.
Time Frame: Predose to 24 hours postdose
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Healthy Controls to Panel A | Panel C: Moderate Renal Impairment | Panel D: Healthy Controls to Panel C | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel H: Healthy Controls to Panel G
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
mL/min | 99.4 (29.1) | 144 (21.9) | 59.6 (29.4) | 136 (23.9) | 24.5 (50.5) | 140 (24.4) | 146 (18.6)

22. Secondary Outcome: Part 2: Plasma AUC0-∞ of Caffeine as a Probe Substrate of Cytochrome P450 Enzyme (CYP)1A2
Description: Caffeine was selected as a substrate of CYP1A2. AUC0-∞ was determined in participants with severe renal impairment and ESRD/HD participants.
Time Frame: Predose and 0.5, 1, 2,3, 4, 8, 12, and 24 hours postdose
Population: Treated participants with severe renal deficiency or ESRD and their matched controls (Panels E-H) who complied with the protocol enough to ensure that generated data were likely to exhibit the effects of treatment, according to the underlying scientific model, are included. Per protocol, Panels A-D were not included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: µM*hr
Groups:
- Panel E: Severe Renal Impairment: Participants with an eGFR <30 mL/min/1.73m² receive an oral cocktail containing caffeine 200 mg, midazolam 2 mg, and omeprazole 40 mg in Part 2.
- Panel G: ESRD/HD Period 1 Postdialysis: Participants with ESRD/HD receive an oral cocktail containing caffeine 200 mg, midazolam 2 mg, and omeprazole 40 mg 1 hour predialysis (Period 1) in Part 2.
- Panel G: ESRD/HD Period 2 Predialysis: Participants with ESRD/HD receive an oral cocktail containing caffeine 200 mg, midazolam 2 mg, and omeprazole 40 mg 24 hours predialysis (Period 2) in Part 2.
Arm/Group | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel G: ESRD/HD Period 2 Predialysis | Panel H: Healthy Controls to Panel G
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
µM*hr | 336 [232 to 489] | 221 [156 to 314] | 190 [138 to 264] | 200 [144 to 277] | 300 [211 to 427]
Statistical Analysis 1: Comparison: Panel E: Severe Renal Impairment vs Panel F: Healthy Controls to Panel E; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 1.52, 90% CI 2-sided [1.07 to 2.15]
Statistical Analysis 2: Comparison: Panel G: ESRD/HD Period 1 Postdialysis vs Panel H: Healthy Controls to Panel G; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.63, 90% CI 2-sided [0.45 to 0.90]
Statistical Analysis 3: Comparison: Panel G: ESRD/HD Period 2 Predialysis vs Panel H: Healthy Controls to Panel G; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.67, 90% CI 2-sided [0.47 to 0.94]

23. Secondary Outcome: Part 2: Plasma AUC0-∞ of Midazolam as a Probe Substrate of Cytochrome P450 Enzyme (CYP)3A4
Description: Midazolam was selected as a substrate of CYP3A4. AUC0-∞ was determined in participants with severe renal impairment and ESRD/HD participants.
Time Frame: Predose and 0.5, 1, 2,3, 4, 8, 12, and 24 hours postdose
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel G: ESRD/HD Period 2 Predialysis | Panel H: Healthy Controls to Panel G
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
µM*hr | 0.130 [0.0730 to 0.230] | 0.121 [0.0707 to 0.207] | 0.0681 [0.0413 to 0.112] | 0.0700 [0.0425 to 0.115] | 0.114 [0.0664 to 0.197]
Statistical Analysis 1: Comparison: Panel E: Severe Renal Impairment vs Panel F: Healthy Controls to Panel E; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 1.07, 90% CI 2-sided [0.63 to 1.83]
Statistical Analysis 2: Comparison: Panel G: ESRD/HD Period 1 Postdialysis vs Panel H: Healthy Controls to Panel G; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.60, 90% CI 2-sided [0.35 to 1.01]
Statistical Analysis 3: Comparison: Panel G: ESRD/HD Period 2 Predialysis vs Panel H: Healthy Controls to Panel G; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.61, 90% CI 2-sided [0.36 to 1.04]

24. Secondary Outcome: Part 2: Plasma AUC0-∞ of Omeprazole as a Probe Substrate of Cytochrome P450 Enzyme (CYP)2C19
Description: Omeprazole was selected as a substrate of CYP2C19. AUC0-∞ was determined in participants with severe renal impairment and ESRD/HD participants.
Time Frame: Predose and 0.5, 1, 2,3, 4, 8, 12, and 24 hours postdose
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Panel E: Severe Renal Impairment | Panel F: Healthy Controls to Panel E | Panel G: ESRD/HD Period 1 Postdialysis | Panel G: ESRD/HD Period 2 Predialysis | Panel H: Healthy Controls to Panel G
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 5
µM*hr | 9.10 [3.34 to 24.8] | 6.20 [2.85 to 13.5] | 4.56 [2.16 to 9.59] | 4.08 [1.97 to 8.44] | 5.03 [2.18 to 11.6]
Statistical Analysis 1: Comparison: Panel E: Severe Renal Impairment vs Panel F: Healthy Controls to Panel E; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 1.47, 90% CI 2-sided [0.63 to 3.40]
Statistical Analysis 2: Comparison: Panel G: ESRD/HD Period 1 Postdialysis vs Panel H: Healthy Controls to Panel G; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.91, 90% CI 2-sided [0.41 to 2.00]
Statistical Analysis 3: Comparison: Panel G: ESRD/HD Period 2 Predialysis vs Panel H: Healthy Controls to Panel G; Test type: Other — GMR (Renal Impairment/Healthy Control); GMR = 0.81, 90% CI 2-sided [0.37 to 1.78]

25. Secondary Outcome: Parts 1 and 2: Percentage of Participants With ≥1 Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 14 days after the last dose of study drug in Part 2 (up to 11 weeks)
Population: All enrolled participants are included in the safety analysis according to the treatment received. Per protocol, healthy matched controls were pooled for the purpose of the safety analysis.
Measure: Number; unit: Percentage of Participants
Groups:
- Panel G: ESRD/HD Participants: Participants with ESRD/HD receive a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV postdialysis (Period 1) and predialysis (Period 2) in Part 1.
- Healthy Matched Controls (Part 1): Healthy matched controls receive a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV. Data from all of the Healthy Control subsets from Part 1 was pooled for safety analyses.
- Panel E: Severe Renal Impairment (Part 2): Participants with Participants with an eGFR <30 mL/min/1.73m² receive an oral cocktail containing caffeine 200 mg, midazolam 2 mg, and omeprazole 40 mg postdialysis (Period 1) and predialysis (Period 2) in Part 2.
- Panel G: ESRD/HD (Part 2): Participants with ESRD/HD receive an oral cocktail containing caffeine 200 mg, midazolam 2 mg, and omeprazole 40 mg postdialysis (Period 1) and predialysis (Period 2) in Part 2.
- Healthy Matched Controls (Part 2): Healthy matched controls receive an oral cocktail containing caffeine 200 mg, midazolam 2 mg, and omeprazole 40 mg postdialysis (Period 1) and predialysis (Period 2) in Part 2. Data from all of the Healthy Control subsets from Part 2 was pooled for safety analyses.
Arm/Group | Panel A: Mild Renal Impairment | Panel C: Moderate Renal Impairment | Panel E: Severe Renal Impairment | Panel G: ESRD/HD Participants | Healthy Matched Controls (Part 1) | Panel E: Severe Renal Impairment (Part 2) | Panel G: ESRD/HD (Part 2) | Healthy Matched Controls (Part 2)
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 24 | 6 | 6 | 12
Percentage of Participants | 28.6 | 16.7 | 16.7 | 33.3 | 0.0 | 33.3 | 33.3 | 0.0

26. Primary Outcome: Dialysis Clearance (CLD) of MK-7655 in Participants With End-stage Renal Diseases Requiring Hemodialysis (ESRD/HD)
Description: The CLD of MK-7655 was determined in ESRD/HD participants for 4.5 hours during HD. The formula for calculating CLD was: CLd = (1-Hct)*QB*[(pre-dialyzer concentration - post-dialyzer concentration) / (pre-dialyzer concentration)] where QB=350 mL/min and Hct=hematocrit.
Time Frame: 1, 1.5, 2, 2.5, 3, 3.5, 4, and 4.5 hours postdose
Population: Treated participants who complied with the protocol sufficiently to ensure that generated data were likely to exhibit the effects of treatment, according to the underlying scientific model, are included. Per protocol, only Panel G participants requiring HD were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Panel G: ESRD/HD Period 2 Predialysis
Number analyzed (Participants) | 6
mL/min
  1 hour postdose: number analyzed (Participants) | 3
  1 hour postdose | 172 (3.5)
  1.5 hours postdose: number analyzed (Participants) | 3
  1.5 hours postdose | 158 (9.4)
  2 hours postdose: number analyzed (Participants) | 4
  2 hours postdose | 170 (5.9)
  2.5 hours postdose: number analyzed (Participants) | 4
  2.5 hours postdose | 166 (7.0)
  3.0 hours postdose | 171 (5.4)
  3.5 hours postdose | 177 (15.7)
  4 hours postdose | 204 (20.2)
  4.5 hours postdose | 198 (23.0)

27. Primary Outcome: Extraction Coefficient of MK-7655 in Participants With End-stage Renal Diseases Requiring Hemodialysis (ESRD/HD)
Description: The extraction coefficient of MK-7655 was determined in ESRD/HD participants for 4.5 hours during HD. The formula for calculating extraction coefficient was: Extraction Coefficient = ABS[100*(post-dialyzer concentration - pre-dialyzer concentration) / pre-dialyzer concentration].
Time Frame: 1, 1.5, 2, 2.5, 3, 3.5, 4, and 4.5 hours postdose
Population: Treated participants who complied with the protocol sufficiently to ensure that generated data were likely to exhibit the effects of treatment, according to the underlying scientific model, are included. Per protocol, only Panel G is included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Extraction coefficient
Arm/Group | Panel G: ESRD/HD Period 2 Predialysis
Number analyzed (Participants) | 6
Extraction coefficient
  1 hour postdose: number analyzed (Participants) | 3
  1 hour postdose | 73 (1.8)
  1.5 hours postdose: number analyzed (Participants) | 3
  1.5 hours postdose | 67 (9.5)
  2 hours postdose: number analyzed (Participants) | 4
  2 hours postdose | 73 (4.5)
  2.5 hours postdose: number analyzed (Participants) | 4
  2.5 hours postdose | 71 (5.6)
  3.0 hours postdose | 73 (4.1)
  3.5 hours postdose | 76 (15.7)
  4 hours postdose | 87 (19.6)
  4.5 hours postdose | 84 (22.2)

ADVERSE EVENTS:
Time Frame: Up to 14 days after the last dose of study drug in Part 2 (up to 11 weeks)
Description: All enrolled participants are included in the safety analysis according to the treatment received. Per protocol, healthy matched controls were pooled for the purpose of the safety analysis. AEs were reported separately for Panels E, G, and matching controls during Parts 1 and 2.
Groups:
- Healthy Matched Controls: Healthy matched controls receive a single dose of MK-7655 125 mg + PRIMAXIN® 250 mg IV in Part 1. For AE reporting, all healthy control participants in Part 1 are pooled into a single arm.
- Panel E: Severe Renal Impairment (Part 2): Participants with an eGFR <30 mL/min/1.73m² receive an oral cocktail containing caffeine 200 mg, midazolam 2 mg, and omeprazole 40 mg.
- Panel G: ESRD/HC (Part 2): Participants with ESRD/HD receive an oral cocktail containing caffeine 200 mg, midazolam 2 mg, and omeprazole 40 mg.
- Healthy Matched Controls (Part 2): Healthy matched controls receive an oral cocktail containing caffeine 200 mg, midazolam 2 mg, and omeprazole 40 mg in Part 2. For AE reporting, all healthy control participants in Part 2 are pooled into a single arm.
Arm/Group | Panel A: Mild Renal Impairment | Panel C: Moderate Renal Impairment | Panel E: Severe Renal Impairment | Panel G: ESRD/HD Participants | Healthy Matched Controls | Panel E: Severe Renal Impairment (Part 2) | Panel G: ESRD/HC (Part 2) | Healthy Matched Controls (Part 2)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/6 | 0/24 | 0/6 | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/6 | 0/24 | 0/6 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 2/7 | 1/6 | 1/6 | 2/6 | 0/24 | 2/6 | 2/6 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panel A: Mild Renal Impairment (N=7) | Panel C: Moderate Renal Impairment (N=6) | Panel E: Severe Renal Impairment (N=6) | Panel G: ESRD/HD Participants (N=6) | Healthy Matched Controls (N=24) | Panel E: Severe Renal Impairment (Part 2) (N=6) | Panel G: ESRD/HC (Part 2) (N=6) | Healthy Matched Controls (Part 2) (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion site swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.